CLINICAL TRIAL: NCT05914740
Title: Feasibility Study of Ultrasound-guided Functional Remodeling of Lower Extremity Superficial Venous Valve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2022110
Record Dates: First submitted 2023-05-24; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Varicose Veins of Lower Limb
Keywords: Varicose veins in the lower extremities; Ultrasonic guidance; venous valve of Lower limb

STUDY DESIGN:
Intervention Model Description: A certain number of patients meeting the requirements (meeting the inclusion criteria, but not meeting the exclusion criteria) were selected for preoperative hemodynamic evaluation of lower extremity vein ultrasound to determine the reflux points and reflux points, identify the blood circulation pattern, and design an individualized surgical program. Intraoperative venous valve was reconstructed in situ under ultrasound guidance. Postoperative ultrasound was used to assess venous valve function and complications in the operative area.
Masking Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venous valve remodeling (Experimental): Venous valve function was remodeled under ultrasound guidance
  Interventions: Procedure: Ultrasound guided functional remodeling of lower extremity superficial vein valve

INTERVENTIONS:
Procedure: Ultrasound guided functional remodeling of lower extremity superficial vein valve — Preoperative ultrasound was used to re-evaluate and confirm the valve function, disinfect the tissue, inject hyaluronic acid around the great saphenous vein valve to reshape the valve about 1-2ml, monitor the whole process under ultrasound, pump back for protection during injection, and inject multiple times at different points.

SUMMARY:
In this project, an exploratory study was conducted to perform in situ venous valve remodeling in vivo, evaluate venous valve function after surgery and conduct regular follow-up, collect relevant ultrasonic data before, during and after surgery, and evaluate the safety and effectiveness of Ultrasound-guided percutaneous great saphenous vein valve functional remodeling.

DETAILED DESCRIPTION:
A certain number of patients meeting the requirements (meeting the inclusion criteria, but not meeting the exclusion criteria) were selected for preoperative hemodynamic evaluation of lower extremity vein ultrasound to determine the reflux points and reflux points, identify the blood circulation pattern, and design an individualized surgical program. Intraoperative venous valve was remodeled in situ under ultrasound guidance. Postoperative ultrasound was used to assess venous valve function and complications in the operative area.

Screening period (before surgery 14 days to 0 days) Subject signs informed consent. General information and previous medical history of subjects were collected, preoperative laboratory examination (blood routine, blood biochemistry, coagulation function, preoperative immunity, blood type), electrocardiogram, ultrasound, preoperative hemodynamic evaluation of lower extremity vein were completed, and evaluation scales such as CEAP grading, VCSS, AVVQ, CIVIQ and pain score were completed.

Subjects who meet the inclusion criteria and do not meet all exclusion criteria will be admitted.

Day of surgery (day 0) Preoperative ultrasound was re-evaluated to confirm the valve function, and the tissue was disinfected. Hyaluronic acid was injected around the valve of the great saphenous vein to rebuild the valve about 1-2ml, and the whole process was monitored under ultrasound. During the injection, the valve function was pumped back for protection, and the injection was performed multiple times at different points. Supplementary injection: Following the subject's voluntary principle, the researcher can give supplementary injection after evaluating the general condition of the subject.

The follow-up period for each subject was 12 months ±20 days after enrollment. Follow-up period (±3 days at 1 week, ±5 days at 1 month, ±10 days at 3 months, ±15 days at 6 months, ±20 days at 1 year) General data of subjects were collected, laboratory examination (blood routine and blood biochemistry) and postoperative ultrasound hemodynamic evaluation of lower limb veins were improved, and evaluation scales such as VCSS, AVVQ, CIVIQ and pain score were completed.

This study does not involve vulnerable groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80, gender unlimited
* CEAP grading was C2-C5 patients
* The patient was clinically diagnosed as a primary varicose great saphenous vein of lower extremity, and the ultrasound findings were great saphenous vein valve insufficiency (complete structure, normal shape, enlarged valve ring, Duration of reflux >0.5s), only unilateral varicose great saphenous vein was treated this time

Exclusion Criteria:

* Patients with target vessel diameter < 3mm
* The final valve of the great saphenous vein was not clear or lost its normal shape on ultrasound
* Patients with deep vein valvular insufficiency
* The presence of thrombus or thrombophlebitis in the main trunk of great cryptic skin
* Target diseased blood vessel had previously received surgical treatment
* Patients with deep vein thrombosis or history of pulmonary distension embolism
* Patients with active implants such as pacemakers or ICDs
* Patients with severe abnormal liver and kidney function (more than three times the normal value)
* Patients with non-primary varicose veins caused by post-deep vein thrombosis syndrome, Cockett syndrome (iliac vein compression syndrome), KT syndrome (venous malformation hypertrophy syndrome >, arteriovenous sputum, etc
* Any serious or uncontrolled systemic disease (including poorly medicated hypertension, diabetes, and diseases with active bleeding signs or severe coagulopathy)
* Patients with diseases that may make treatment and evaluation difficult (e.g., malignant arsine tumor, acute infectious diseases, sepsis, systemic intolerability of surgery, life expectancy less than 12 months, etc.)
* Pregnant and lactating women, or those who planned to have children during the study period
* Patients who have participated in clinical trials of other drugs or medical devices within the last 3 months
* Anesthetist and other patients were deemed unsuitable for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Venous valve regurgitation or not | immediately after intervention
  Under the calf compression test, the venous valves were observed for blood flow regurgitation signal
Venous valve regurgitation or not | 1 week after intervention
  Under the calf compression test, the venous valves were observed for blood flow regurgitation signal
Venous valve regurgitation or not | 1 month after intervention
  Under the calf compression test, the venous valves were observed for blood flow regurgitation signal
Venous valve regurgitation or not | 3 months after intervention
  Under the calf compression test, the venous valves were observed for blood flow regurgitation signal
Venous valve regurgitation or not | 6 months after intervention
  Under the calf compression test, the venous valves were observed for blood flow regurgitation signal
Venous valve regurgitation or not | 1 year after intervention
  Under the calf compression test, the venous valves were observed for blood flow regurgitation signal
Changes in the duration of venous valve regurgitation | immediately after intervention
  The duration of venous valve regurgitation was measured under calf compression test
Changes in the duration of venous valve regurgitation | 1 week after intervention
  The duration of venous valve regurgitation was measured under calf compression test
Changes in the duration of venous valve regurgitation | 1 month after intervention
  The duration of venous valve regurgitation was measured under calf compression test
Changes in the duration of venous valve regurgitation | 3 months after intervention
  The duration of venous valve regurgitation was measured under calf compression test
Changes in the duration of venous valve regurgitation | 6 months after intervention
  The duration of venous valve regurgitation was measured under calf compression test
Changes in the duration of venous valve regurgitation | 1 year after intervention
  The duration of venous valve regurgitation was measured under calf compression test

CONTACTS AND LOCATIONS:
Overall Officials: Yuefeng Zhu, Master's, Study Director — The Fourth Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang Procince, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Maeseneer MG, Kakkos SK, Aherne T, Baekgaard N, Black S, Blomgren L, Giannoukas A, Gohel M, de Graaf R, Hamel-Desnos C, Jawien A, Jaworucka-Kaczorowska A, Lattimer CR, Mosti G, Noppeney T, van Rijn MJ, Stansby G, Esvs Guidelines Committee, Kolh P, Bastos Goncalves F, Chakfe N, Coscas R, de Borst GJ, Dias NV, Hinchliffe RJ, Koncar IB, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, Bjorck M, Labropoulos N, Lurie F, Mansilha A, Nyamekye IK, Ramirez Ortega M, Ulloa JH, Urbanek T, van Rij AM, Vuylsteke ME. Editor's Choice - European Society for Vascular Surgery (ESVS) 2022 Clinical Practice Guidelines on the Management of Chronic Venous Disease of the Lower Limbs. Eur J Vasc Endovasc Surg. 2022 Feb;63(2):184-267. doi: 10.1016/j.ejvs.2021.12.024. Epub 2022 Jan 11. No abstract available. PMID 35027279
- [Result] Muhlberger D, Brenner E, Frings N, Geier B, Mumme A, Reich-Schupke S, Steffen HP, Stenger D, Stucker M, Hummel T. Functional repair of the great saphenous vein by external valvuloplasty reduces the vein's diameter: 6-month results of a multicentre study. J Int Med Res. 2021 May;49(5):3000605211014364. doi: 10.1177/03000605211014364. PMID 33990156